CLINICAL TRIAL: NCT06287684
Title: Molecular Subtype-Specific Mechanisms and Therapeutic Strategies in Sepsis
Acronym: MENDSEP
Status: Recruiting | Type: Observational
Sponsor: Mater Dei Hospital, Malta (Other)
Collaborators: University of Malta (Other)
Responsible Party: Principal Investigator, Brendon Scicluna, PhD, Assistant Professor and Principal Investigator, Mater Dei Hospital, Malta
Other Study IDs: SINO-MALTA-2024-40; ESICM-22
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Bronchoalveolar lavage fluid (BAL), whole blood, Paxgene blood, plasma, and serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Sepsis (all-cause): Suspected infection accompanied by organ dysfunction identified as a total SOFA score ≥ 2 points diagnosed within 24 hours after ITU admission. Definition in line with the Sepsis-3 criteria.
- Non-infectious critical illness: Patients admitted to the ITU with non-infectious etiologies, including trauma.
- Control subjects: Age-, sex-, and comorbidity-matched participants from the community or long term care facility

SUMMARY:
Sepsis is a complex syndrome that causes lethal organ dysfunction due to an abnormal host response to infection. No drug specifically targeting sepsis has been approved. The heterogeneity in sepsis pathophysiology hinders the identification of patients who would benefit, or be harmed, from specific therapeutic interventions. Recent clinical genomics studies have shown that sepsis patients can be stratified as molecular subtypes, or subclasses, with clinical implications. Classifying sepsis patients as molecular subtypes revealed that a poor prognosis subtype was characterized by immunosuppression and septic shock. Therefore, it has become essential to identify patients who may benefit from or be adversely affected by specific treatments, thereby identifying bona fide treatable traits or endotypes. The goal of this study is to assist the physician at the bedside in tailoring the treatment of an individual patient suffering from sepsis by generating rapid molecular information about immune status.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Consent card signed

Exclusion criteria:

* Consent card not signed
* Pregnancy
* Prisoners
* Elective cardiac surgery patients with an uncomplicated stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All-cause sepsis, non-infectious critical illness, and control participants
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Molecular subtype assignments | Through study completion, an average of 2 year
  Molecular subtype classification of sepsis patients using a consensus transcriptomic subtype model
Molecular information about the host response in patients with sepsis | Through study completion, an average of 2 year
  Measurement of soluble mediators of host immune responses, including inflammation, coagulation, endothelial function

SECONDARY OUTCOMES:
Survival | 3 years
  Assessment of survival

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Dei hospital, Intensive Therapy Unit, Msida, Malta

IPD SHARING:
Plan to Share IPD: No